CLINICAL TRIAL: NCT01709331
Title: A Phase III, Multi-center, Open Label, Uncontrolled Trial to Investigate the Efficacy and Safety of MK-8962 (Corifollitropin Alfa) in Combination With Human Chorionic Gonadotropin (hCG) in Inducing Increased Testicular Volume and Spermatogenesis in Adult Men With Hypogonadotropic Hypogonadism Who Remain Azoospermic When Treated With hCG Alone (Phase III; Protocol No. MK-8962-031-00 [Also Known as SCH 900962, P07937])
Brief Title: A Study of the Efficacy and Safety of Corifollitropin Alfa (MK-8962) in Combination With Human Chorionic Gonadotropin (hCG) in Adult Men With Hypogonadotropic Hypogonadism (HH) (P07937)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P07937; 2012-001258-25 (EudraCT Number); MK-8962-031 (Other: Merck)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Hypogonadism; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corifollitropin alfa 150 μg + hCG (Experimental): During a 16-week pretreatment phase, participants will receive twice-weekly subcutaneous (SC) injections of hCG 1500 or 3000 international units (IU). Eligible participants will then be enrolled in the combined treatment phase in which they will receive a single dose of corifollitropin alfa 150 μg by SC injection once every 2 weeks for 52 weeks. In addition, eligible participants will continue to receive twice-weekly hCG injections on the same schedule as the pretreatment phase.
  Interventions: Drug: Corifollitropin alfa; Drug: hCG

INTERVENTIONS:
Drug: Corifollitropin alfa — Corifollitropin alfa 150 μg by SC injection, once every 2 weeks for 52 weeks
  Other Names: MK-8962
Drug: hCG — hCG 1500 or 3000 IU by SC injection twice a week; administered alone for 16 weeks (pre-treatment phase) and then in combination with corifollitropin alfa for 52 weeks (combined treatment phase)

SUMMARY:
This study will assess if corifollitropin alfa (MK-8962), when administered in combination with human chorionic gonadotropin (hCG), will increase testicular volume in men with HH who remain azoospermic after treatment with hCG alone.

Hypothesis: The lower limit of the 95% confidence interval for the geometric mean increase in testicular volume from Day 1 to Week 52 is greater than one.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypogonadotropic hypogonadism, either congenital or acquired
* Have low circulating levels of testosterone
* Have low circulating levels of gonadotropins (follicle stimulating hormone [FSH]; luteinizing hormone)
* Presence of both scrotal testes
* Have azoospermia (no measurable level of sperm)
* Adequate replacement of other pituitary hormones
* Good general physical and mental health

Exclusion Criteria:

* Primary hypogonadism, such as Klinefelter's syndrome
* History of unilateral or bilateral cryptorchidism (maldescended testes)
* History or presence of testicular pathology of clinical importance (e.g., epididymitis, orchitis, testicular torsion, varicocele stage III, testicular atrophy, occlusive azoospermia, etc), and/or vasectomy
* Treated with FSH, hCG or gonadotropin-releasing hormone (GnRH) within previous 3 months or for more than 1 month within previous 6 months
* Proven spermatogenesis with hCG treatment alone
* Previous unsuccessful attempt with hCG in combination with human menopausal gonadotropin (hMG)/FSH to achieve spermatogenesis
* Required a dose of hCG of more than 6000 international units (IU) per week in a previous attempt to normalize T levels
* Untreated pituitary or hypothalamic tumor, or inadequately treated pituitary or hypothalamic tumor that is likely to progress during the study
* History or presence (known or suspected) of testicular, prostatic or breast cancer
* Prostate pathology of clinical importance
* Past or present oncologic treatment (chemo/radiotherapy)
* Diabetes mellitus
* Clinically significant, untreated hyperprolactinaemia
* Uncontrolled non-gonadal endocrinopathies (thyroid, adrenal, pituitary disorders)
* Tested positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
* User of recreational or illicit drugs or has had a recent history (within the past year) of drug abuse or dependence, or increased alcohol consumption
* Allergy/sensitivity to gonadotropins or its/their excipients
* Has received within previous 1 month or plans to use: Hormonal preparations other than the study medication, drugs that are known to impair testicular function, agents known to affect sex hormone secretion and/or drugs that are known or suspected to be teratogenic
* Used any investigational drugs within three months or actively participating in another study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2015-04-08 (Actual); Study Completion 2015-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nieschlag E, Bouloux PG, Stegmann BJ, Shankar RR, Guan Y, Tzontcheva A, McCrary Sisk C, Behre HM. An open-label clinical trial to investigate the efficacy and safety of corifollitropin alfa combined with hCG in adult men with hypogonadotropic hypogonadism. Reprod Biol Endocrinol. 2017 Mar 7;15(1):17. doi: 10.1186/s12958-017-0232-y. PMID 28270212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-three participants entered the 16-week pretreatment phase with hCG. At the end of the pretreatment phase, 18 participants were enrolled in the 52-week combined treatment phase.
Groups:
- Corifollitropin Alfa 150 μg + hCG: During a 16-week pretreatment phase, participants received twice-weekly subcutaneous (SC) injections of human chorionic gonadotropin (hCG) 1500 or 3000 IU. Eligible participants were then enrolled in the combined treatment phase in which they received a single dose of corifollitropin alfa 150 μg by SC injection once every 2 weeks for 52 weeks. In addition, eligible participants continued to receive twice-weekly hCG injections on the same schedule begun during the pretreatment phase.
Period: Overall Study
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the combined treatment phase
Groups:
- Corifollitropin Alfa 150 μg + hCG: During a 16-week pretreatment phase, participants received twice-weekly SC injections of hCG 1500 or 3000 IU. Eligible participants were then enrolled in the combined treatment phase in which they received a single dose of corifollitropin alfa 150 μg by SC injection once every 2 weeks for 52 weeks. In addition, eligible participants continued to receive twice-weekly hCG injections on the same schedule begun during the pretreatment phase.
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log-Transformed Testicular Volume at Week 52
Description: Participants underwent testicular ultrasound in the pretreatment phase at Weeks -16, -8, -1; and during the combined treatment phase at Baseline (predose, Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52. The testicular volume was measured as the sum of volumes of left and right testes. The mean change from Day 1 in log-transformed testicular volume was analyzed using a mixed model with a fixed effect for time point and a random effect for the participant. For each time point, the mean change from Day 1 to that time point and the associated 95% confidence interval (CI) was calculated. The geometric mean fold change in testicular volume and its 95% CI was obtained by exponentiation.
Time Frame: Baseline and Week 52
Population: Full Analysis Set (FAS) population, which consisted of all participants who received any dose of corifollitropin alfa and who had a baseline and at least one post-baseline measurement of testicular volume.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Number analyzed (Participants) | 18
Fold change | 2.3 [2.03 to 2.62]

2. Primary Outcome: Percentage of Participants With Anti-Corifollitropin Alfa Antibodies
Description: Blood samples were collected for assessment of anti-corifollitropin alfa antibodies in the pretreatment phase at Week -16 and Week -1; during the combined treatment phase at Weeks 4, 16, 28, 50, 52; and at the post-treatment follow-up visit, which could occur from Week 53 up to Week 57.
Time Frame: Up to Week 57
Population: All-Subjects-as-Treated (ASaT) population, which consisted of all participants who received any dose of corifollitropin alfa.
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Number analyzed (Participants) | 18
Percentage of participants | 0 [52.4 to 93.6]

3. Secondary Outcome: Percentage of Participants With Induced Spermatogenesis Resulting in a Sperm Count ≥1x10^6/mL at or Before Week 52
Description: Semen samples were produced by masturbation after at least 48 hours of sexual abstinence and collected for evaluation in the pretreatment phase at Week -1, and during the combined treatment phase at Weeks 16, 28, 40, and 52.
Time Frame: Up to Week 52
Population: FAS population, which consisted of all participants who received any dose of corifollitropin alfa and who had a baseline and at least one post-baseline measurement of testicular volume.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Number analyzed (Participants) | 18
Percentage of participants | 77.8 [52.4 to 93.6]

ADVERSE EVENTS:
Time Frame: Up to Week 57
Description: The Safety Analysis was based on the ASaT population, which consisted of all participants who received any dose of corifollitropin alfa.
Arm/Group | Corifollitropin Alfa 150 μg + hCG
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 150 μg + hCG (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (5)
Blood pressure increased (Investigations) | 1 (1)
Blood testosterone increased (Investigations) | 2 (2)
Oestradiol increased (Investigations) | 3 (4)
Testicular scan abnormal (Investigations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Blood testosterone decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, e.g., any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.